CLINICAL TRIAL: NCT02864238
Title: The Utility of an Electronic Based Milestone Pathway on the Care of Patients Undergoing Cardiac Valve Surgery
Brief Title: The Utility of Clinical Milestones Pathway in a Cardiovascular ICU
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Adam Kingeter, Assistant Professor, Vanderbilt University
Other Study IDs: IRB #151566
Record Dates: First submitted 2016-07-13; First posted 2016-08-11 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Cardiac Surgery
Keywords: electronic milestone pathway; cardiac valve surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre intervention: This cohort consists of patients who underwent cardiac valve surgery during calender year 2013 prior to the institution of the electronic milestone pathway
- post intervention: This cohort consists of patients who underwent cardiac valve surgery during calender year 2014 after the electronic milestone pathway had been instituted
  Interventions: Other: electronic milestone pathway

INTERVENTIONS:
Other: electronic milestone pathway — an electronic based, clinical milestone driven pathway developed to guide the care of cardiac valve surgery patients.
  Groups: post intervention

SUMMARY:
The economic burden of health care is becoming a greater burden from year to year. Medicare spending, which represented 20 percent of national health spending in 2013, grew 3.4 percent to $585.7 billion, a slowdown from growth of 4.0 percent in 2012. This slowdown was attributed largely to slower enrollment growth and impacts of the Affordable Care Act (ACA) and sequestration. Per-enrollee spending in 2013 grew at about the same rate as 2012.

The push to create Accountable Care Organizations (ACO) has taken these initiatives a step further. The goal would be to move away from a fee for service system and base reimbursement on quality of care. Clinical metrics, re-admissions, and patient satisfaction in categories of acute myocardial infarction, congestive heart failure, pneumonia, surgeries and healthcare associated infections will be the foci for 2013. Centers for Medicare and Medicaid Services (CMS) has also initiated a valve bundled payment system that encompasses total patient care for 90 days, including readmissions.

Leapfrog and the ACO movement along with the nonprofit group Institute for Health Care Improvement have placed quality and cost effectiveness into the spotlight for clinicians in the ICU and beyond. While clinicians have always been focused on evidence based therapies with little concern for cost, in the new era of healthcare understanding cost, value and effectiveness of therapies will be key for improved patient outcomes and institutional solvency in trying economic times.

Vanderbilt elected to enroll in the CMS valve bundle trial. The Leadership team in the heart and vascular institute identified the importance of an electronic medical record that includes display and utilization of key drivers of quality and success across the continuum of care (Preoperative assessment to discharge up to 90 days) in the bundled payment model of care. A multidisciplinary team was developed in conjunction with nurses, midlevel providers, multi-specialty physicians, case managers, informatics specialists, and performance improvement representatives to develop an electronic pathway of care using evidence based and best practices for cardiac surgery.

DETAILED DESCRIPTION:
A multidisciplinary team consisting of physicians, pharmacists, nutritionists, social workers, bedside nurses, physical therapists, and mid-level providers developed the structure and key elements of the milestone pathway. The Vanderbilt University Informatics Team developed the electronic version of the consensus milestones. The pathway encompasses 17 phases beginning with the pre-procedure evaluation and continuing through the perioperative period until the three-month follow-up post procedure. The nursing staff performed documentation of pathway stages during the index hospitalization, and the milestone stage was displayed on the door of the patient's room. The milestone stage was discussed on multi-disciplinary bedside rounds in the ICU, and if a patient could not progress to the next stage the nurse would document the reason for failure to progress.

In this study, the investigators compared patients who underwent valve surgery with the milestone pathway in place, to patients who underwent valve surgery without the milestone pathway in place. Patients were adjusted according to baseline characteristics such as demographics, procedure, and proceduralist collected from the electronic medical record and Society of Thoracic Surgeons (STS) database.

The investigators primary clinical outcome is mortality, and secondary clinical outcomes include the incidence of re-intubation within 48 hours, acute kidney injury as defined by Kidney Disease Improving Global Outcome (KDIGO) criteria, delirium, major adverse cardiac events (MACE), and infection rates for catheter and central line associated infections as well as sternal wound infection. In addition the investigators examined financial outcomes including variance in direct and total cost, and direct and total cost per patient.

ELIGIBILITY:
Inclusion Criteria:

* Underwent cardiac valve surgery at vanderbilt university medical center between 1/1/2013 and 12/31/2014

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent cardiac valve surgery at vanderbilt university medical center between 1/1/2013 and 12/31/2014
Sampling Method: Non-Probability Sample
Enrollment: 2401 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
mortality | Post operative day 0 to post operative day 7
  mortality rate for patients during index hospitalization

SECONDARY OUTCOMES:
Re-intubation rate within 48 hours | 48 hours of index procedure
  re-intubation rate within 48 hours of index procedure for patients undergoing cardiac surgery
Acute Kidney Injury as defined by KDIGO (Kidney Disease Improving Global Outcomes) guidelines | All time points occurring between post operative day 0 and Post operative day 7
  Incidence of acute Kidney Injury as defined by KDIGO (Kidney Disease Improving Global Outcomes) guidelines during index hospitalization
Delirium | All time points occurring between post operative day 0 and Post operative day 7
  Incidence of delirium as defined by Intensive Care Unit Confusion Assessment Method (ICU-CAM) scoring system during index hospitalization
major adverse cardiac events | All time points occurring between post operative day 0 and Post operative day 7
  Incidence of major adverse cardiac events defined as death, need for re-operation, myocardial infarction during index hospitalization
Infection rates | All time points occurring between post operative day 0 and Post operative day 7
  defined as Catheter Associated Urinary Tract Infection (CAUTI), Central Line Associated Blood Stream Infection (CLABSI), sternal wound infection during index hospitalization
Direct cost | All time points occurring between post operative day 0 and Post operative day 7
  summation of costs directly attributable to patient care during index hospitalization
total cost | All time points occurring between post operative day 0 and Post operative day 7
  summation of costs directly attributable to patient care, as well as costs to the patient which are not directly attributable to patient care (unspecified charges to patient such as OR utilization fees, laboratory staff fees, etc.)
variance in cost | All time points occurring between post operative day 0 and Post operative day 7
  total and direct costs attributable to each patient undergoing cardiac valve surgery will be averaged for all patients undergoing cardiac valve surgery during the study period. Each individual patient's direct and total costs will then be compared to the averaged cost for all patients undergoing cardiac valve surgery hospitalization to obtain a variance in cost for each individual patient undergoing cardiac valve surgery. The investigators will then compare average variance between the two cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Parmley, MD, JD, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No